CLINICAL TRIAL: NCT05236777
Title: Long-term Surveillance of Patients With Multiple Sclerosis to Report Progressive Multifocal Leukoencephalopathy and Other Serious Opportunistic Infections Among Patients Treated With Natalizumab
Brief Title: TOPIK Study: A Study to Report Progressive Multifocal Leukoencephalopathy and Other Serious Opportunistic Infections in Natalizumab Treated Participants
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Collaborators: ReMuS Registry (Unknown)
Responsible Party: Sponsor
Other Study IDs: CZ-TYS-12155
Record Dates: First submitted 2022-02-02; First posted 2022-02-11 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Multiple Sclerosis
Keywords: Progressive Multifocal Leukoencephalopathy (PML)
MeSH Terms: conditions — Multiple Sclerosis; Leukoencephalopathy, Progressive Multifocal | interventions — Natalizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Natalizumab Cohort: The cohort will include participants with MS who are newly treated with natalizumab (administered as a standard of care/routine clinical practice) from 1st January 2019 including those participants who terminate or discontinue the treatment during the observational period.
  Interventions: Drug: Natalizumab

INTERVENTIONS:
Drug: Natalizumab — Administered as specified in the treatment arm.
  Other Names: Tysabri

SUMMARY:
The primary objective of the study is to estimate the incidence of progressive multifocal leukoencephalopathy (PML) and serious adverse events (SAEs) of other opportunistic infections (OIs) among all participants taking natalizumab. The secondary objectives of the study are to estimate the incidence of SAEs, to estimate the incidence of SAEs among participant subgroups defined by demographic and clinical factors (age, gender, duration of treatment, pregnancy, breastfeeding), to characterize and estimate incidences of malignancies, hypersensitivity reactions and John Cunningham Virus (JCV) positivity among all participants taking natalizumab, and to count and describe pregnancies and breastfeeding among participants previously exposed to natalizumab.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants starting with natalizumab after 1st January 2019 and participating in the ReMuS will be included in this study

Key Exclusion Criteria:

* Not Applicable (NA)

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include participants with MS who are treated with natalizumab from the 1st of January 2019 and participating in the Czech National MS registry (ReMuS).
Sampling Method: Non-Probability Sample
Enrollment: 675 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Progressive Multifocal Leukoencephalopathy (PML) who are Taking Natalizumab | Up to 6 years
Number of Participants with Serious Adverse Events (SAEs) of Other Opportunistic Infections (OIs) who are Taking Natalizumab | Up to 6 years
  SAE means such adverse event that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in permanent or significant damage to health or limitation of capabilities or is manifested as a congenital anomaly or birth defect in offspring, irrespective of the administered dose of the medicinal product. Serious OI means such OI which results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in permanent or significant damage to health or limitation of capabilities or is manifested as a birth defect in offspring.

SECONDARY OUTCOMES:
Number of Participants With SAEs | Up to 6 years
  SAE means such adverse event that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in permanent or significant damage to health or limitation of capabilities or is manifested as a congenital anomaly or birth defect in offspring, irrespective of the administered dose of the medicinal product.
Number of Participants With SAEs Among Participant Subgroups Defined by Demographic and Clinical Factors | Up to 6 years
  SAE means such adverse event that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in permanent or significant damage to health or limitation of capabilities or is manifested as a congenital anomaly or birth defect in offspring, irrespective of the administered dose of the medicinal product. Demographic and clinical factors involve age, gender, duration of treatment, pregnancy, breastfeeding.
Number of Participants With Malignancies who are Taking Natalizumab | Up to 6 years
Number of Participants With Hypersensitivity Reactions who are Taking Natalizumab | Up to 6 years
Number of Participants who are John Cunningham Virus (JCV) Positive and Taking Natalizumab | Up to 6 years
Number of Pregnant and Breastfeeding Participants who Were Previously Exposed to Natalizumab | Up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (15):
- Czechia (15):
  - Fakultní nemocnice Brno, Brno
  - Fakultní nemocnice u sv. Anny v Brně, Brno
  - Nemocnice České Budějovice, České Budějovice
  - Fakultní nemocnice Hradec Králové, Hradec Králové
  - Nemocnice Jihlava, Jihlava
  - Fakultní nemocnice Olomouc, Olomouc
  - Fakultní nemocnice v Ostravě, Ostrava
  - Nemocnice Pardubického kraje, Pardubice
  - Fakultní nemocnice v Plzni, Pilsen
  - Fakultní nemocnice Královské Vinohrady v Praze, Prague
  - Fakultní nemocniceMotol v Praze, Prague
  - Fakultní Thomayerova nemocnice v Praze v Krči, Prague
  - Všeobecná fakultní nemocnice v Praze, Prague
  - Nemocnice Teplice, Teplice
  - Krajská nemocnice T. Bati ve Zlíně, Zlín

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/